CLINICAL TRIAL: NCT06060574
Title: Effect of the Menstrual Cycle on Levels of Growth Factors From Platelet-rich Fibrin and the Size Outcomes of Membrane
Brief Title: Menstrual Cycle and Platelet-rich Fibrin
Status: Not yet recruiting | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Zeynep Tastan Eroglu, assistant professor, Necmettin Erbakan University
Other Study IDs: PRFzeynep
Record Dates: First submitted 2023-09-01; First posted 2023-09-29 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Menstrual Cycle
Keywords: Menstrual cycle; growth factor; Platelet-rich fibrin; hematological parameters; phases of menstrual cycle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The demographic data of the individuals included in the study will be recorded. The MC 1-2 of each individual in the study. days, 8-10. on days (PF), 12-14. days (OD) and premenstrual (PmD) 22-24. 2 tubes of blood samples, approximately 10 ml, will be taken from each individual on the following days. The blood samples taken will be used to create PRF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Menstrual Cycle 1-2nd days: The Blood samples will be drawn from the participants on 1st-2nd day of the menstrual cycle of each of these 36 participants. PRF will be obtained from the blood taken these days.
  Interventions: Device: Platelet rich fibrin device
- Menstrual Cycle 8-10. days : proliferative phase (PP): The Blood samples will be drawn from the participants on 8-10. days of the menstrual cycle of each of these 36 participants. PRF will be obtained from the blood taken these days.
  Interventions: Device: Platelet rich fibrin device
- Menstrual Cycle 12-14. days: ovulation phase (OP): The Blood samples will be drawn from the participants on 12-14. days of the menstrual cycle of each of these 36 participants. PRF will be obtained from the blood taken these days.
  Interventions: Device: Platelet rich fibrin device
- premenstrual (PmD) 22-24. days: The Blood samples will be drawn from the participants on 22-24. days of the menstrual cycle of each of these 36 participants. PRF will be obtained from the blood taken these days.
  Interventions: Device: Platelet rich fibrin device

INTERVENTIONS:
Device: Platelet rich fibrin device — Within the scope of the study, a total of 2 tubes of venous blood samples will be obtained from the forearm region (antecubital vein) of each individual by the clinical staff specialist nurse of the Department of Periodontology. PRF samples will be created using appropriate equipment and devices from blood samples obtained from each individual. In the study, 10 ml glass-coated plastic tubes will be used. Apart from this, 5 mL of blood taken will be used for complete blood count and evaluation of hormones on the relevant day.
  PRF Preparation: In all age groups, PRF will be prepared by centrifugation with 700xg (=2700 rpm, Intra-Spin L-PRF device) for 12 minutes.

SUMMARY:
The goal of this clinical trial is to test effect of menstrual cycle (MC) on growth factors of platelet rich fibrin (PRF) in health condition. The main questions it aims to answer are:

question 1: Does MC have an effect on growth factors in PRF? question 2: In which menstrual phase are growth factors higher? question 3:Does the change in the number of blood cells in the menstrual cycle have an effect on PRF? Participants will describe the main tasks participants will be asked to do.

DETAILED DESCRIPTION:
Abstract Platelet-rich fibrin (PRF) is frequently used in periodontal regenerative treatments. Thanks to the growth factors in its content, it affects the healing positively. Studies have shown that the size and content of PRF are affected by variables such as age, gender, centrifugation speed and inflammation.

It is known that during the menstrual cycle (MS) phases in women, changes occur in cell numbers and growth factors in the blood. The aim of this study is to determine the size of the PRF and the epidermal growth factor (EGF), insulin-like growth factor-1 (IGF-1), platelet-derived growth factor-BB (PDGF-BB), transforming growth factor-β1 (TGF-β1) and vascular endothelial growth factor (VEGF).

PRF membrane will be formed from the blood of each individual in the study, taken on days 1-2 (M), 8-10 (PF), 12-14 (OD) and days 22-24 before menstruation (PmD). The size of the membranes will be measured. On the same days, individuals will have a complete blood count. The growth factors levels of each PRF membrane obtained at the 1st, 24th and 72nd hours will be determined.

At the end of the study, the growth factors contents of the PRF membranes obtained in different phases of MS will be compared. In addition, the effect of the results of the complete blood count of the individuals on the PRF membrane will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Having a regular MS in the last three periods and a menstrual period lasting 5-7 days,
* Not using contraceptive drugs and/or drugs that affect sex hormones,
* With less than 10% bleeding on probing within 10 seconds after probing, that is, gingival ally healthy,
* Have not received any periodontal or orthodontic treatment until at least 6 months before the start of the study,
* Have not used antibiotics in the last 6 months for any reason
* Systemically healthy individuals without prosthetic restoration in their mouths will be included.

Exclusion Criteria:

* Those who have any systemic disease and drug use related to it
* Pregnant or breastfeeding
* have recently used aspirin or have a disease related to the clotting process
* Refusing to participate in the study

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Erbakan University Faculty of Dentistry who meet the following inclusion criteria will be included in the study. Eligibility of the individuals to be included in the study. Instructor It will be evaluated at NEU Faculty of Dentistry Periodontology Clinic.
  The sample size of the study was calculated with the help of R Statistical Language (version 4.1.2; The R Foundation for Statistical Computing, Vienna, Austria; http://www.r-project.org). In order to determine whether there is a significant difference between the 4 different mestural phases of women in terms of growth factor levels, it was planned to perform the study with at least 36 individuals with 5% significance level, 95% statistical power and 0.25 effect size for Variance analysis in Repeated Measurements.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-11-28 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in EGF in the obtained PRF during the menstrual cycle | 1 month
  PRF membrane will be formed from the blood of each individual in the study, taken on days 1-2 (M), 8-10 (PF), 12-14 (OD) and days 22-24 before menstruation (PmD). EGF levels of each PRF membrane obtained at the 1st, 24th and 72nd hours will be determined.
  At the end of the study, EGF contents of the PRF membranes obtained in different phases of MS will be compared.
Changes in IGF-1 in the obtained PRF during the menstrual cycle | 1 month
  PRF membrane will be formed from the blood of each individual in the study, taken on days 1-2 (M), 8-10 (PF), 12-14 (OD) and days 22-24 before menstruation (PmD). IGF-1 levels of each PRF membrane obtained at the 1st, 24th and 72nd hours will be determined.At the end of the study, IGF-1 contents of the PRF membranes obtained in different phases of MS will be compared.
Changes in PDGF in the obtained PRF during the menstrual cycle | 1 month
  PRF membrane will be formed from the blood of each individual in the study, taken on days 1-2 (M), 8-10 (PF), 12-14 (OD) and days 22-24 before menstruation (PmD). PDGF levels of each PRF membrane obtained at the 1st, 24th and 72nd hours will be determined.
  At the end of the study, PDGF contents of the PRF membranes obtained in different phases of MS will be compared.
Changes in TGF-beta in the obtained PRF during the menstrual cycle | 1 month
  PRF membrane will be formed from the blood of each individual in the study, taken on days 1-2 (M), 8-10 (PF), 12-14 (OD) and days 22-24 before menstruation (PmD). TGF-beta levels of each PRF membrane obtained at the 1st, 24th and 72nd hours will be determined.
  At the end of the study, TGF-beta contents of the PRF membranes obtained in different phases of MS will be compared.
Changes in VEGF in the obtained PRF during the menstrual cycle | 1 month
  PRF membrane will be formed from the blood of each individual in the study, taken on days 1-2 (M), 8-10 (PF), 12-14 (OD) and days 22-24 before menstruation (PmD). VEGF levels of each PRF membrane obtained at the 1st, 24th and 72nd hours will be determined.
  At the end of the study, VEGF contents of the PRF membranes obtained in different phases of MS will be compared.

SECONDARY OUTCOMES:
Change in the proportion of red blood cells and its effect on PRF. | 1 month
  PRF membrane will be formed from the blood of each individual in the study, taken on days 1-2 (M), 8-10 (PF), 12-14 (OD) and days 22-24 before menstruation (PmD).At the same time, complete blood count of the participants will be done. Changes in the proportion of red blood cells throughout MS will be examined. The effect of changes in the proportion of red blood cells on PRF size will be evaluated. PRF length and width will be measured in mm. The proportion of red blood cells will be evaluated with hematocrit level, an instrument for measuring the ratio of the volume of red blood cells to the total volume of blood.